CLINICAL TRIAL: NCT01152697
Title: A Prospective Trial of Customized Adherence Enhancement Plus Long-acting Injectable Antipsychotic (CAE-L) in Individuals With Schizophrenia or Schizoaffective Disorder at Risk for Treatment Non-adherence and for Homelessness
Brief Title: Customized Adherence Enhancement Plus Long-acting Injectable Antipsychotic
Acronym: CAE-L
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Martha Sajatovic, Professor of Psychiatry, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Reuter-L1473
Record Dates: First submitted 2010-06-24; First posted 2010-06-29 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Patient Noncompliance
Keywords: nonadherence; noncompliance; homeless; schizophrenia; schizoaffective
MeSH Terms: conditions — Patient Compliance; Schizophrenia | interventions — haloperidol decanoate; Haloperidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patient Noncompliance (Experimental): There was only one arm for this study.
  Interventions: Drug: haloperidol decanoate; Drug: haloperidol; Behavioral: Customized Adherence Enhancement

INTERVENTIONS:
Drug: haloperidol decanoate — Drug is in in injectable form and will be administered approximately every four weeks through Week 25 of the study. A participant may continue on the drug after Week 25 at the discretion of his or her treating psychiatrist. Dosage is per package insert or at the discretion of the psychiatrist.
Drug: haloperidol — Drug will be administered in oral form to participants not already taking oral haloperidol and then transitioned to the injectable version. Dosage and frequency is at the discretion of the psychiatrist.
Behavioral: Customized Adherence Enhancement — CAE targets key areas relevant to non-adherent populations with schizophrenia or schizoaffective disorder: 1) inadequate or incorrect understanding of mental disorder; 2) lack of medication-taking routines; 3) poor communication with care providers; and 4) substance use which interferes with adherence and healthy behaviors that promote recovery. CAE is delivered based upon initial assessment of reasons for non-adherence and only those components of CAE that are determined to be indicated for that individual are delivered (psychoeducation, modified motivational interviewing, assistance with medication routines, coaching in communication with providers).

SUMMARY:
Psychotropic medications are a cornerstone of treatment for individuals with schizophrenia and schizoaffective disorder, however rates of full or partial non-adherence can exceed 60%. Inadequate adherence is associated with poor outcomes such as relapse, homelessness, hospitalization, and increased health care costs. Studies have shown a direct correlation between non-adherence and rates of relapse in schizophrenia; on average, non-adherent patients have a risk of relapse that is 3.7 times greater than their adherent counterparts. A major obstacle to good outcomes in the maintenance treatment of patients with severe mental illness is difficulty with medication routines on an on-going basis. For this reason, long-acting injectable antipsychotic medication is a particularly attractive treatment option for populations with schizophrenia and schizoaffective disorder, although it is unlikely that medication treatment alone is likely to modify long-term attitudes and behaviors.

This prospective study is a pilot analysis of a combined approach which merges a psychosocial intervention to optimize treatment attitudes towards psychotropic medication (CAE) and long-acting injectable antipsychotic medication (L) in recently homeless individuals with schizophrenia or schizoaffective disorder who are known to have on-going difficulties with treatment non-adherence. It is expected that this combined approach (CAE-L) will improve illness outcomes among the most vulnerable of populations with schizophrenia or schizoaffective disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals age 18 years old and older with schizophrenia or schizoaffective disorder as confirmed by the Mini International Psychiatric Inventory (MINI).
2. Individuals who are currently or have been recently homeless (within the past 12 months) as per the official federal definition of homelessness.
3. Known to have medication treatment adherence (20% or more missed medications in past week or past month) problems as identified by the Treatment Routines Questionnaire patient or clinician versions (TRQ-P/TRQ-C).
4. Ability to be rated on psychiatric rating scales.
5. Willingness to take long-acting injectable medication.
6. Currently receiving treatment at a Community Mental Health Clinic (CMHC) or another mental health treatment provider who is able to provide continuity of care during and after study participation.
7. Able to provide written, informed consent to study participation.
8. Women of child-bearing potential must be utilizing reliable, medically-accepted methods of birth control.

Exclusion Criteria:

1. Known resistance or intolerance to haloperidol or haloperidol decanoate.
2. Medical contraindication to haloperidol or haloperidol decanoate.
3. Individuals on long-acting injectable antipsychotic medication immediately prior to study enrollment.
4. Prior or current treatment with clozapine.
5. Concurrent medical condition or psychiatric illness, which in the opinion of the research psychiatrist, would interfere with the patient's ability to participate in the trial.
6. Current substance dependence.
7. High risk of harm to self or others.
8. Female who is currently pregnant or breastfeeding.
9. Individual who is already in permanent and supported housing that includes comprehensive mental health services (e.g. Housing First).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hosptials, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Sajatovic M, Levin J, Ramirez LF, Hahn DY, Tatsuoka C, Bialko CS, Cassidy KA, Fuentes-Casiano E, Williams TD. Prospective trial of customized adherence enhancement plus long-acting injectable antipsychotic medication in homeless or recently homeless individuals with schizophrenia or schizoaffective disorder. J Clin Psychiatry. 2013 Dec;74(12):1249-55. doi: 10.4088/JCP.12m08331. PMID 24434094

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Noncompliance: Only one arm for this study. Interventions given were as follows: study drugs haloperidol decanoate or haloperidol and behavioral intervention called Customized Adherence Enhancement (CAE). Dosage form was a long acting injectable administered every three to five weeks. Mean endpoint dose was 68.0 mg.
Period: Overall Study
Arm/Group | Patient Noncompliance
Started | 30
Completed | 11
Not Completed | 19

BASELINE CHARACTERISTICS:
Groups:
- Patient Noncompliance: Only one arm for this study. Interventions given were as follows: study drugs haloperidol decanoate or haloperidol and behavioral intervention called Customized Adherence Enhancement (CAE).
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.77 (8.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Days Homeless Out of the Previous 6 Months as Measured at 25 Weeks
Description: Subjects will be asked how many days they have been homeless
Time Frame: Baseline-25 weeks
Population: 26 participants were asked how many days they were homeless at week 25. Only data for these participants was analyzed for change from baseline to week 25.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 26
days
  Baseline | 6.50 (7.73)
  25 Weeks | 9.85 (13.96)

2. Primary Outcome: Change From Baseline in Treatment Adherence Score as Measured at 25 Weeks
Description: A total treatment adherence score will calculated as a proportion of medications taken as reported from the participant, and evidenced by pill counts and documented medication injections.
Time Frame: Baseline-25 weeks
Population: 17 participants were administered and completed measurement of their Treatment Adherence scores at week 25. Only data for these participants was analyzed for change from baseline to week 25.
Measure: Mean (Standard Deviation); unit: Percentage of doses
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 17
Percentage of doses
  Past week | 30.91 (34.50)
  Past month | 10.10 (16.70)

3. Primary Outcome: Change From Baseline in Adherence Attitude Score as Measured by the Drug Attitude Inventory (DAI) at 25 Weeks
Description: Ten item inventory taken by the participant with a Scale Range: 0-10. Higher scores indicate improved outcomes.
Time Frame: Baseline-25 weeks
Population: 15 participants were administered and completed measurement with the DAI at week 25. Only data for these participants was analyzed for change from baseline to week 25.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 15
units on a scale
  Baseline | 7.47 (1.84)
  Week 25 | 8.07 (1.03)

4. Primary Outcome: Change From Baseline in Treatment Adherence Behavior Score as Measured by the Morisky Medication Rating Scale at 25 Weeks
Description: Four item inventory taken by participant with Scale Range: 0-4. Lower scores indicate improved outcomes.
Time Frame: Baseline-25 weeks
Population: 16 participants were administered and completed measurement with the Morisky Medication Rating Scale at week 25. Only data for these participants was analyzed for change from baseline to week 25.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 16
units on a scale
  Baseline | 2.31 (1.20)
  Week 25 | 1.19 (1.47)

5. Primary Outcome: Change From Baseline in Adherence Attitude Score as Measured by the Attitude Toward Medication Questionnaire (AMQ) at 25 Weeks
Description: Nineteen item inventory taken by the participant with Scale Range:0-19. Lower scores indicate improved outcomes.
Time Frame: Baseline-25 weeks
Population: 19 participants were administered and completed measurement with the AMQ at week 25. Only data for these participants was analyzed for change from baseline to week 25. Lower scores indicate improved outcomes.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 19
units on a scale
  Baseline | 6.63 (3.44)
  Week 25 | 4.47 (3.29)

6. Secondary Outcome: Frequency of Health Resource Use Throughout Months 10, 11, and 12
Description: The frequency of health resource use will be measured through interview of the participant.
Time Frame: Month 1-3, Month 10-12
Population: Three participants were administered and completed this measurement at 12 months. Only data for these participants was analyzed for changes.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 3
days
  3 Month | 19.33 (27.65)
  12 Month | 15.50 (20.51)

7. Secondary Outcome: Change in Serious Mental Illness Severity Score as Measured by the Brief Psychiatric Rating Scale (BPRS) at 25 Weeks
Description: The BPRS, developed by Overall and Gorham (1962), is a widely used, relatively brief scale that measures major psychotic and non-psychotic symptoms in individuals with SMI. The 18-item BPRS is well-validated and is perhaps the most researched instrument in psychiatry. Reliability coefficients are reported to be in the range of 0.56-0.87.
  Scale Range: 18-126 Lower scores represent improved outcomes.
Time Frame: Baseline-25 weeks
Population: 19 participants were administered and completed measurement with the BPRS at week 25. Only data for these participants was analyzed for change from baseline to week 25.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 19
units on a scale
  Baseline | 46.37 (9.87)
  Week 25 | 32.84 (10.03)

8. Secondary Outcome: Change in Global Psychopathology as Measured by the Clinical Global Impressions (CGI) at 25 Weeks
Description: Global psychopathology will be measured with the Clinical Global Impressions (CGI) (Guy 1976) a widely used scale which evaluates illness severity on a 1 to 7 point continuum. Severity of illness ratings on the CGI have reported reliability scores ranging from 0.41-0.66 (Guy 1976) Lower scores indicate improved outcomes. Higher scores indicate worse outcomes.
  Illness scale: 1 - 7 (1 = Normal/not at all ill ; 7 = Among the most extremely ill patients) Global improvement scale: 1 - 7 (1 = Very much improved ; 7 = Very much worse)
Time Frame: Baseline-25 weeks
Population: 17 participants were administered and completed measurement with the DAI at week 25. Only data for these participants was analyzed for change at week 25.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 17
units on a scale
  Baseline - Severity | 4.76 (0.83)
  Week 25 - Severity | 3.24 (0.75)
  Baseline - Global Improvement | 3.43 (0.98)
  Week 25 - Global Improvement | 2.14 (0.90)

9. Secondary Outcome: Change in Social and Occupational Functioning Scale (SOFAS) as Measured at 25 Weeks
Description: Life and Work Functional status will be evaluated using the Social and Occupational Functioning Scale (SOFAS), which is derived from the GAF (Global Assessment of Functioning). The GAF is a 100-point single-item scale which measures global functioning of psychiatric patients and is widely utilized in clinical studies involving Seriously Mentally Ill patients (Jones 1995). The reliability of the GAF ranges from 0.62-0.82. Higher scores indicate improved outcomes.
Time Frame: Baseline-25 weeks
Population: 17 participants were administered and completed measurement with the SOFAS at week 25. Only data for these participants was analyzed for change from baseline to week 25.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 17
units on a scale
  Baseline | 47.35 (6.92)
  Week 25 | 58.65 (10.05)

10. Secondary Outcome: Treatment Satisfaction as Measured by the Participant Acceptability and Satisfaction Questionnaire at 25 Weeks
Description: Satisfaction will be measured by a seven item inventory taken by the participant.
  Scale ranges from 1 (Strongly Agree) to 5 (Strongly Disagree). Lower scores indicate better outcomes, while higher scores indicate worse outcomes. The highest possible score is 35.
Time Frame: 25 weeks
Population: 17 participants were administered and completed this measure at week 25.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 17
units on a scale | 12.12 (3.92)

11. Secondary Outcome: Change in Schizophrenia and Schizoaffective Disorder Symptom Severity Scale as Measured by the Positive and Negative Syndrome Scale (PANSS) at 25 Weeks
Description: The PANSS (Kay, Fiszbein, & Opler 1987) was created to assess both the positive and negative symptoms of schizophrenia such as hallucinations and emotional withdrawal, respectively. The scale rates 30 symptoms on a scale from 1 (absent) to 7 (extreme) and has been shown to limit bias between the assessment of positive and negative symptoms, providing a broad but balanced spectrum of the illness.
  There are three subscales: positive symptoms, negative symptoms, general psychopathology. Potential responses to Items on all subscales range from 1 (absent) to 7 (extreme). Lower scores indicate lower symptoms and, therefore, better outcomes. Higher scores indicate more presence of symptoms and, therefore, worse outcomes.
  Subscales are combined to produce a total score, which is summed from all of the subscales. Lower total scores indicate lower symptoms and, therefore, better outcomes. Higher total scores indicate more presence of symptoms and, therefore, worse outcomes.
Time Frame: Baseline-25 weeks
Population: 19 participants were administered and completed measurement with the PANSS at week 25. Only data for these participants was analyzed for change from baseline to week 25.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 19
units on a scale
  Baseline | 46.37 (9.87)
  Week 25 | 32.84 (10.03)

12. Secondary Outcome: Frequency of Health Resource Use in the Past 3 Months as Measured at 25 Weeks
Description: The frequency of health resource use will be measured through interview of the participant.
Time Frame: 25 weeks
Population: 17 participants were administered and completed this measure at week 25.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 17
days | 20.18 (35.92)

13. Secondary Outcome: Global Psychopathology as Measured by the Clinical Global Impressions (CGI) at 12 Months
Description: as for outcome 8
Time Frame: 12 months
Population: 12 participants were administered and completed measurement with the CGI at 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 12
units on a scale
  Severity | 3.17 (0.84)
  Global Improvement | 2.42 (0.90)

14. Secondary Outcome: Change in Social and Occupational Functioning Scale (SOFAS) as Measured at 12 Months
Description: Life and Work Functional status will be evaluated using the Social and Occupational Functioning Scale (SOFAS), which is derived from the GAF. The GAF is a 100-point single-item scale which measures global functioning of psychiatric patients and is widely utilized in clinical studies involving Seriously Mentally Ill patients (Jones 1995). The reliability of the GAF ranges from 0.62-0.82. Higher scores indicate improved outcomes.
Time Frame: Baseline-12 months
Population: Six participants were administered and completed measurement with the SOFAS at 12 months. Only data for these participants was analyzed for change from baseline to 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 6
units on a scale
  Baseline | 45.33 (5.13)
  12 months | 63.83 (10.53)

15. Secondary Outcome: Treatment Satisfaction as Measured by the Participant Acceptability and Satisfaction Questionnaire at 12 Months
Description: as for outcome 10
Time Frame: 12 months
Population: Six participants were administered and completed this measure at 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 6
units on a scale | 12.33 (2.50)

16. Secondary Outcome: Days Homeless Out of the Previous 6 Months as Measured at 12 Months
Description: Subjects will be asked how many days they have been homeless
Time Frame: 12 months
Population: Six participants were administered and completed this measure at 12 months.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 5
days | 35 (47.96)

17. Secondary Outcome: Treatment Adherence Score as Measured at 12 Months
Description: as for outcome 2
Time Frame: 12 months
Population: Seven participants were administered and completed this measure at 12 months.
Measure: Mean (Standard Deviation); unit: Percentage of doses
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 7
Percentage of doses
  Past Week | 28.65 (34.03)
  Past Month | 6 (7.48)

18. Secondary Outcome: Adherence Attitude Score as Measured by the Drug Attitude Inventory (DAI) at 12 Months
Description: Ten item inventory taken by the participant with a Scale Range: 0-10. Higher scores indicate improved outcomes.
Time Frame: 12 months
Population: Six participants were administered and completed this measure at 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 6
units on a scale | 7.00 (1.67)

19. Secondary Outcome: Treatment Adherence Behavior Score as Measured by the Morisky Medication Rating Scale at 12 Months
Description: Four item inventory taken by participant with Scale Range: 0-4. Lower scores indicate better outcomes.
Time Frame: 12 months
Population: Six participants were administered and completed this measure at 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 6
units on a scale | 1.33 (1.03)

20. Secondary Outcome: Adherence Attitude Score as Measured by the Attitude Toward Medication Questionnaire (AMQ) at 12 Months
Description: Nineteen item inventory taken by the participant with Scale Range:0-19. Lower scores indicate improved outcomes.
Time Frame: 12 months
Population: Seven participants were administered and completed this measure at 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Noncompliance
Number analyzed (Participants) | 7
units on a scale | 2.43 (1.27)

ADVERSE EVENTS:
Arm/Group | Patient Noncompliance
Serious Adverse Events (participants affected / at risk) | 6/30
Other Adverse Events (participants affected / at risk) | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient Noncompliance (N=30)
Abnormal EKG (Cardiac disorders) | 1 (1) — Not due to cardiac condition or study drug, as reviewed by the cardiologist.
Stomach Cramps (Gastrointestinal disorders) | 1 (1)
High Blood Pressure (Cardiac disorders) | 1 (1) — Patient was already prescribed blood pressure medication and had not yet started taking study drug at the time of the incident.
Toothache and Infection (Infections and infestations) | 1 (1)
Infection in Leg (Infections and infestations) | 1 (1)
Complications from Colostomy Surgery (Infections and infestations) | 1 (2) — Infection from surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No